CLINICAL TRIAL: NCT01914848
Title: Multiprofessional Advance Care Planning and Shared Decision-making for End of Life Care MAPS Trial
Brief Title: Multiprofessional Advance Care Planning and Shared Decision Making for End of Life Care
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MAPS Trial
Record Dates: First submitted 2012-11-26; First posted 2013-08-02 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Palliative Patients; Surrogate Decision Maker
MeSH Terms: interventions — Advance Care Planning; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): A routine care discharge planning with the social service
  Interventions: Other: Control Group
- Advance Care Planning ACP (Experimental): Patient get a decision aid video and library and up to 3 consultations with qualified Advance Care Planning Facilitators.
  --------------------------------------------------------------------------------
  Interventions: Other: Advance Care Planning ACP

INTERVENTIONS:
Other: Advance Care Planning ACP — Patient of the intervention group get a decision aid video and library and up to 3 consultations with qualified Advance Care Planning Facilitators.
  Arms: Advance Care Planning ACP
Other: Control Group — A routine care discharge planning with the social service
  Arms: Control Group

SUMMARY:
Multiprofessional Advance Care Planning and shared decision making for end of live care for terminal patients and their relatives.

The aim of this study is to develop, implement and test a complex intervention for improving patients' preparation for and participation in end of life decisions. In cooperation with local, national and international partners, the investigators will focus on strategies to enhance advance care planning and shared decision making on end of life issues, and documentation and transferability of end of life decisions across health care settings in coordinated approach involving patients, their families and care givers (in and out of hospital).

ELIGIBILITY:
Inclusion criteria: -patients in which the treating physician on the ward would not be surprised if the patient died during the next year (surprise question of Weissman et al 2011)

* male and female patients above 18 years of age
* signed informed consent after being informed
* patients able to appoint a surrogate decision maker (SM) and/or responsible physician to be contacted after discharge

Exclusion criteria: -patients not capable of speaking german

* patients having no responsible physician to be contacted after discharge and no relative/future surrogate decision maker (SM)
* inhouse patients being discharged within the next 2 days or ambulatory patients not regularly coming to the wards (at least every two month)
* patients assessed by their physician to be in obvious denial of their situation (illness/prognosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
end of life wish on resuscitation known (if alive) or fulfilled(if dead) after 6 month by responsible physician and/or surrogate decision maker (SM) | during 2 weeks six months after discharge

SECONDARY OUTCOMES:
end of live decisions on last place of care, antibiotics for pneumonia, feeding tube, intravenous fluids, dialysis, intubation and sedation, | during 2 weeks six months after discharge
decisional conflict scale ("DCS"), O Connor et al 1995 | at discharge and during 2 Weeks six months after discharge
Satisfaction with information and care, (see Detering et al 2010) | at discharge
Hospital Anxiety and Depression scale ("HADS") | discharge and during 2 weeks six months after discharge
Having an Advance directive | at discharge, during 2 weeks three months after discharge and during 2 weeks six months after discharge
Having an appointed surrogate decision maker | at discharge, during 2 weeks three month after discharge and during 2 weeks six month after discharge
Any hospital stay | during 2 weeks three months after discharge and during 2 weeks six months after discharge
Decisions regarding end of life issues already having been made/taken place | during 2 weeks six months after discharge
open question on important medical decisions being made | during 2 weeks three months after discharge
Treatment against patients wishes | during 2 weeks three months after discharge and during 2 weeks six months after discharge, or 3 month after death
Distress of Patients or relatives because of content of the consultation | at discharge, during 2 weeks three months after discharge and during 2 weeks six months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Krones, MD, Principal Investigator — University Hospital Zurich, Clinical Ethics
Locations (1):
- University Hospital Zurich, Clinical Ethics, Zurich, Canton of Zurich, Switzerland